CLINICAL TRIAL: NCT04607733
Title: A Bioequivalence Study of Injections of Mirikizumab Solution Using an Investigational 1-mL Pre-Filled Syringe and an Investigational 1-mL Autoinjector in Healthy Participants
Brief Title: A Study of Mirikizumab in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17820; I6T-MC-AMBW (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-10-28; First posted 2020-10-29 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mirikizumab - Prefilled Syringe (Experimental): 2× 1mL (total 200 milligrams (mg) mirikizumab) administered by subcutaneous injection (SC) via a prefilled syringe (PFS)
  Interventions: Drug: Mirikizumab Prefilled Syringe
- Mirikizumab - Autoinjector (Experimental): 2× 1mL (total 200 milligrams (mg) mirikizumab) administered by subcutaneous injection (SC) via an autoinjector (AI)
  Interventions: Drug: Mirikizumab Autoinjector

INTERVENTIONS:
Drug: Mirikizumab Prefilled Syringe — Administered SC by prefilled syringe
  Other Names: LY3074828
  Arms: Mirikizumab - Prefilled Syringe
Drug: Mirikizumab Autoinjector — Administered SC by autoinjector
  Other Names: LY3074828
  Arms: Mirikizumab - Autoinjector

SUMMARY:
The main purpose of this study is to compare the amount of mirikizumab that gets into the blood stream and how long it takes the body to get rid of it, when given as a solution formulation via manual prefilled syringe or autoinjector. The information about any adverse effects experienced will be collected and the tolerability of mirikizumab will also be evaluated.

Screening is required within 28 days prior to the start of the study. For each participant, the total duration of the clinical trial will be about 17 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined through medical history and physical examination

Exclusion Criteria:

* Must not have an average weekly alcohol intake that exceeds 21 units/week (males) and 14 units/week (females)
* Must not show evidence of active or latent tuberculosis (TB)
* Must not have received live vaccine(s) (including attenuated live vaccines and those administered intranasally) within 8 weeks of screening, or intend to during the study
* Must not have been treated with steroids within 1 month of screening, or intend to during the study
* Must not be immunocompromised
* Must not have received treatment with biologic agents (e.g. monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to Day 1
* Must not have clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or severe post treatment hypersensitivity reactions
* Must not have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Must not have had breast cancer within the past 10 years
* Must not have significant allergies to humanized monoclonal antibodies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Covance Clinical Research Inc, Daytona Beach, Florida
  - QPS, Springfield, Missouri
  - Covance Dallas, Dallas, Texas
  - Covance Clinical Research Inc, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Otani Y, Payne CD, Morris NJ, Chua L, Escobar R, Wang S, Shi G. Pharmacokinetic Bridging Between an Autoinjector and a Prefilled Syringe Following Subcutaneous Administration of Mirikizumab in Healthy Participants. Adv Ther. 2025 Nov;42(11):5529-5546. doi: 10.1007/s12325-025-03335-z. Epub 2025 Sep 3. PMID 40900263

RESULTS

PARTICIPANT FLOW:
Groups:
- AI (Test) Abdomen: AI (Test) Abdomen:
  2× 1mL (total 200 milligrams (mg) mirikizumab) administered by subcutaneous injection (SC) via an autoinjector (AI).
- AI (Test) Arm: AI (Test) Arm:
  2× 1mL (total 200 mg mirikizumab) administered by subcutaneous injection (SC) via an autoinjector (AI).
- AI (Test) Thigh: AI (Test) Thigh:
  2× 1mL (total 200 mg mirikizumab) administered by subcutaneous injection (SC) via an autoinjector (AI).
- PFS (Reference) Abdomen: PFS (Reference) Abdomen:
  2× 1mL (total 200 mg mirikizumab) administered by subcutaneous injection (SC) via a prefilled syringe (PFS).
- PFS (Reference) Arm: PFS (Reference) Arm:
  2× 1mL (total 200 mg mirikizumab) administered by subcutaneous injection (SC) via a prefilled syringe (PFS).
- PFS (Reference) Thigh: PFS (Reference) Thigh:
  2× 1mL (total 200 mg mirikizumab) administered by subcutaneous injection (SC) via a prefilled syringe (PFS).
Period: Overall Study
Arm/Group | AI (Test) Abdomen | AI (Test) Arm | AI (Test) Thigh | PFS (Reference) Abdomen | PFS (Reference) Arm | PFS (Reference) Thigh
Started | 40 | 39 | 41 | 40 | 41 | 39
Received at Least One Dose of Drug | 40 | 39 | 41 | 40 | 41 | 39
Completed | 39 | 39 | 41 | 39 | 39 | 39
Not Completed | 1 | 0 | 0 | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- AI (Test): AI (Test):
  2× 1mL (total 200 mg mirikizumab) administered by subcutaneous injection (SC) via an autoinjector (AI).
- PFS (Reference): PFS (Reference):
  2× 1mL (total 200 mg mirikizumab) administered by subcutaneous injection (SC) via a prefilled syringe (PFS).
- Total: Total of all reporting groups
Arm/Group | AI (Test) | PFS (Reference) | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.0) | 40.1 (12.4) | 41.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 71 | 139
  Male | 52 | 49 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 20 | 41
  Not Hispanic or Latino | 99 | 100 | 199
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 19 | 30 | 49
  White | 97 | 83 | 180
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 120 | 120 | 240

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Mirikizumab
Description: PK: Cmax of Mirikizumab
Time Frame: Predose up to 85 days postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data for this outcome.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/mL)
Arm/Group | PFS (Reference) | AI (Test)
Number analyzed (Participants) | 120 | 120
micrograms/milliliter (µg/mL) | 14.3 (44) | 15.2 (40)

2. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Mirikizumab
Description: PK: AUC[0-∞] of Mirikizumab
Time Frame: Predose up to 85 days postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*day/milliliter (µg*day/mL)
Arm/Group | PFS (Reference) | AI (Test)
Number analyzed (Participants) | 120 | 120
micrograms*day/milliliter (µg*day/mL) | 246 (44) | 262 (39)

3. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Measured Concentration Value (AUC[0-tlast]) of Mirikizumab
Description: PK: AUC[0-tlast] of Mirikizumab
Time Frame: Predose up to 85 days postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*day/milliliter (µg*day/mL)
Arm/Group | PFS (Reference) | AI (Test)
Number analyzed (Participants) | 116 | 119
micrograms*day/milliliter (µg*day/mL) | 244 (44) | 257 (39)

ADVERSE EVENTS:
Time Frame: Baseline Up To 85 Days
Description: All participants who received at least one dose of study drug.
Groups:
- AI (Test) Abdomen: AI (Test) Abdomen:
  2× 1mL (total 200 mg mirikizumab) administered by subcutaneous injection (SC) via an autoinjector (AI).
Arm/Group | AI (Test) Abdomen | AI (Test) Arm | AI (Test) Thigh | PFS (Reference) Abdomen | PFS (Reference) Arm | PFS (Reference) Thigh
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39 | 0/41 | 0/40 | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39 | 0/41 | 0/40 | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 7/40 | 6/39 | 8/41 | 6/40 | 5/41 | 6/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AI (Test) Abdomen (N=40) | AI (Test) Arm (N=39) | AI (Test) Thigh (N=41) | PFS (Reference) Abdomen (N=40) | PFS (Reference) Arm (N=41) | PFS (Reference) Thigh (N=39)
Injection site reaction (General disorders) | 3 (6) | 3 (5) | 4 (8) | 2 (4) | 4 (8) | 3 (5)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 4 (5) | 3 (3) | 4 (4) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT04607733/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT04607733/SAP_001.pdf